CLINICAL TRIAL: NCT02922114
Title: Comparison of the Clinical Examination and the Joint Ultrasonography in the Evaluation of Disease Activity in Systemic Lupus Patients
Brief Title: Comparison of the Clinical Examination and the Joint Ultrasonography in Lupus Patients
Acronym: LUPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2013-02
Record Dates: First submitted 2016-09-27; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Ultrasonography; Clinical assesment; joint abnormalities
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasonography (Experimental): B-mode and power Doppler Ultrasonography examination
  Interventions: Other: Ultrasonography

INTERVENTIONS:
Other: Ultrasonography — B-mode and power Doppler ultrasonography examination.Ultrasonography assessments includes wrists, metacarpophalangeal, proximal interphalangeal, elbows, shoulders, knees, ankles, metatarsophalangeal and twenty six tendons (wrist extensors, finger flectors and tendons of the ankles).

SUMMARY:
Arthritis is a current manifestation of systemic lupus erythematosus (SLE) and participates to the SLEDAI composite score calculation (0 to 105). Ultrasonography (US) is a validated and sensitive tool for joint assessment. Published studies showed US joint abnormalities in systemic lupus erythematosus patients with or without joint pain. Nevertheless, ultrasonography evaluations were not standardized and no study compared clinical and ultrasonography assessments. The objectives were 1) to describe ultrasonography joint abnormalities in systemic lupus erythematosus population, 2) to compare clinical and ultrasonography standardized joint assessments, 3) to estimate the reliability of clinical swollen joint count (C-SJC) and SLEDAI (C-SLEDAI) score versus ultrasonography-SJC and ultrasonography-SLEDAI.

ELIGIBILITY:
Inclusion Criteria:

* Systemic Lupus Erythematosus patients (with or without joint involvement).
* subjects will have to sign the inform consent before the beginning of the study

Exclusion Criteria:

* Current pregnancy or no effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Ultrasonography record (synovitis / tenosynovitis / effusion) | Day 0 (there is only one point measurement in the study)
Clinical joint assessment (synovitis / tenosynovitis / effusion) | Day 0
Evaluate SELENA SLEDAI (C-SLEDAI) score | Day 0
Evaluate musculoskeletal BILAG score | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Carine SALLIOT, Principal Investigator — CHR ORLEANS
Locations (7):
- France (7):
  - Hopital Pellegrin, Bordeaux
  - Chu de Brest, Brest
  - CH du MANS, Le Mans
  - CHU Hôtel Dieu, Nantes
  - CHR d'Orléans, Orléans La Source
  - Hopital Pontchaillon - Chu de Rennes, Rennes
  - Chru de Tours, Tours

IPD SHARING:
Plan to Share IPD: No